CLINICAL TRIAL: NCT07069296
Title: Impact of Gestational Diabetes on Childhood Obesity and Related Metabolic Disorders in Children Aged 5-12
Brief Title: Impact of Gestational Diabetes on Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Gul, Prof Dr Ali Gul, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022/59
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gestatiaonl Diabetes Mellitus; Insulin Resistance; Dyslipaemia; Obesity &Amp; Overweight
Keywords: Obesity; children; gestational diabetes mellitus; insulin resistance; dyslipidemia
MeSH Terms: conditions — Insulin Resistance; Obesity; Overweight; Diabetes, Gestational; Dyslipidemias | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children aged 5 to 12 years, born to mothers without a diagnosis of GDM (Placebo Comparator): Control
  Interventions: Diagnostic Test: blood samples were collected from participants; Diagnostic Test: blood samples
- children aged 5 to 12 years, born to mothers with a diagnosis of GDM (Active Comparator): Patient group
  Interventions: Diagnostic Test: blood samples were collected from participants; Diagnostic Test: blood samples

INTERVENTIONS:
Diagnostic Test: blood samples were collected from participants — Blood samples obtained
Diagnostic Test: blood samples — Blood sampling

SUMMARY:
In this study, we aimed to investigate the relationship between obesity, glucose intolerance (insulin resistance), dyslipidemia and diabetes in children aged 5-12 born to mothers with Gestational Diabetes Mellitus (GDM) in Gaziosmanpaşa University Hospitals in Tokat province. The effect of GDM on both obesity and obesity-related disorders was examined.

DETAILED DESCRIPTION:
Patients diagnosed with gestational diabetes mellitus (GDM) were identified through the automation system of Gaziosmanpaşa University Faculty of Medicine. Patient records were reviewed retrospectively, and the patients were contacted by phone to provide detailed information about the study. Children eligible for inclusion were invited to the hospital, and informed consent was obtained from their parents.

Patients presenting to the outpatient clinic were evaluated for obesity. Data including sex, gestational age at birth, birth weight, breastfeeding status, height, and body weight were recorded. Height and weight percentiles, body mass index (BMI), and Z-scores were calculated using the automated program available on the website of the Turkish Pediatric Endocrinology Society (https://www.ceddcozum.com/).

During height measurements, children were instructed to remove their shoes and stand upright against a flat wall so that the back of their head, shoulders, hips, and heels touched the wall. A stadiometer was used to perform the measurement. Body weight was measured using a precise digital scale while the children wore light clothing and no shoes. Based on their percentiles, children were categorized as underweight, normal weight, overweight, or obese. A BMI at or above the 95th percentile was classified as "obese," between the 85th and 94th percentile as "overweight," between the 5th and 84th percentile as "normal weight," and below the 5th percentile as "underweight" (40, 41). The study group included those with a BMI between the 5th and 85th percentile (BMI-SDS between -1 and +1), while the obese group consisted of those at or above the 95th percentile (BMI-SDS +2 and above) (42).

Fasting blood samples were drawn after an 8-hour fasting period. From all children, laboratory tests including total cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL), very low-density lipoprotein (VLDL), high-density lipoprotein (HDL), fasting insulin, glucose, electrolytes (Na, K, Cl), blood urea nitrogen (BUN), creatinine, complete blood count, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) levels were analyzed. After obtaining the results, the homeostatic model assessment of insulin resistance (HOMA-IR) was calculated using the following formula:

HOMA-IR = [fasting insulin (mIU/ml) × fasting glucose (mg/dl)] / 405. Insulin resistance in children was determined based on HOMA-IR values. In prepubertal children, values above 2.67 for boys and 2.22 for girls were considered positive. In pubertal children, values above 5.22 for boys and 3.82 for girls were considered positive (43).

For the control group, healthy children aged 5-12 years without any chronic illness or endocrinological disorder, who presented to the pediatric outpatient clinic at Gaziosmanpaşa University Faculty of Medicine Hospital, were included. Informed consent was obtained from their parents. Sex, gestational age, birth weight, breastfeeding status, height, weight, and BMI were recorded, and blood tests were performed.

An application for funding support was submitted to the Scientific Research Projects Coordination Unit of Gaziosmanpaşa University. The project was approved for funding on 31.05.2022.

Ethical approval was obtained from the Tokat Gaziosmanpaşa University Clinical Research Ethics Committee (Approval Number: 22-KAEK-10). Additionally, permission was obtained from the hospital administration to access and use the hospital automation system.

Patients with congenital heart disease were excluded from the study. A total of 35 children born to mothers with gestational diabetes were identified. One child was excluded due to congenital heart disease, and the study was conducted with 34 children. A total of 40 healthy children were included in the control group. Children with chronic diseases such as hypothyroidism, familial hyperlipidemia, or diabetes were excluded from the control group.

Descriptive statistics were used to summarize the general characteristics of the study groups. Continuous variables were expressed as mean ± standard deviation (SD), and categorical variables as n (%). The significance of differences between group means for continuous variables was assessed using the Independent Samples t-test. Relationships between categorical variables were examined using cross-tabulations and Chi-square tests. Pearson correlation coefficients were used to assess relationships between continuous variables. A p-value of <0.05 was considered statistically significant. Statistical analyses were performed using SPSS version 19.0 (Chicago, IL, USA)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years, born to mothers diagnosed with GDM, were included in the study The control group consisted of children aged 5-12 years, recruited from a pediatric outpatient clinic, who had no history of maternal GDM

Exclusion Criteria:

* Chi,ldren had chronic illnesses, or endocrinological disorders

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Obesity frequency | 1 to 2 year
  This study aimed to evaluate the incidence of obesity in children aged 5-12 years born to mothers with GDM and to examine the role of GDM in the development of obesity

SECONDARY OUTCOMES:
obesity-related metabolic disorders | 1 to 2 year
  Fasting blood samples were collected to analyze serum insulin levels, lipid profiles, thyroid function tests, fasting glucose. The homeostasis model assessment of insulin resistance (HOMA-IR) was calculated using the following formula: HOMA-IR = [fasting insulin (mIU/mL) × fasting glucose (mg/dL)]/405 (12, 13). Insulin resistance (IR) was defined as a HOMA-IR value greater than 2.67 in prepubertal boys, 2.22 in prepubertal girls, 5.22 in pubertal boys, and 3.82 in pubertal girls

CONTACTS AND LOCATIONS:
Overall Officials: Ali Gul, Professor, Study Chair — Tokat Gaziosmanpasa University
Locations (1):
- Clinic of Pediatrics, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Concept - AG, EA; Design - AG, EA; Supervision - AG, TK, ST; Funding - AG, EK; Materials - EA, AG; Data Collection and/or Processing - EA, AG, EK; Analysis and/or Interpretation: AG, EA, TK, Writing - AG, EA; Critical Review - TK, ST.
Time Frame: May 15 2022